CLINICAL TRIAL: NCT01202214
Title: A Randomized, Single-Blind, Placebo Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GSK1440115 After a Single Dose and 7 Days of Repeat Dosing in Healthy Volunteers
Brief Title: Repeat Dose Safety Study for Compound to Treat Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Accenture (Industry)
Responsible Party: Nancy Smerkanich, Vice President, Regulatory Affairs, Octagon Research Solutions, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UR2114661
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — 4'-(1-(((6,7-dichloro-3- oxo-2,3-dihydro-4H-1,4-benzoxazin-4-yl)acetyl)(methyl)amino)-2-(4-morpholinyl)ethyl)-4-biphenylcarboxylic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active drug (Experimental)
  Interventions: Drug: 1440115
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1440115
  Arms: Active drug
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to describe the safety and tolerability of single and repeat oral doses of GSK1440115 in healthy volunteers.

DETAILED DESCRIPTION:
This study is the first administration of GSK1440115 to humans. GSK1440115 is a urotensin II receptor antagonist which is being developed for the treatment of asthma. This will be a two-part study to evaluate the safety, tolerability, and pharmacokinetics of single (Part A) and repeat (Part B) oral doses of GSK1440115 in healthy adult male and female (of non-child bearing potential) subjects. This study will be a randomized, single-blind, placebo-controlled, dose escalation design. Part A will evaluate a single dose of GSK1440115. Part B will evaluate repeat daily doses for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
2. Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
3. A female subject is eligible to participate if she is of:

   - Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
4. Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study drug until completion of the Follow-up Period.
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
6. AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
7. QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening
2. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
3. A positive pre-study drug/alcohol screen.
4. A positive test for HIV antibody.
5. Average systolic blood pressure of < 100 mmHg at Screening.
6. History of regular alcohol consumption within 6 months of the study defined as:

   - an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
8. Use of prescription or non-prescription medications, vitamins, and dietary or herbal supplements (including St John's Wort) within 7 days (or 14 days if the medication is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
9. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
10. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
11. Pregnant females as determined by positive serum or urine hCG test at Screening or prior to dosing.
12. Lactating females.
13. Unwillingness or inability to follow the procedures outlined in the protocol.
14. Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2010-09

PRIMARY OUTCOMES:
Safety and tolerability assessments consisting of Adverse Events, ECGs, vital signs, clinical observations, and clinical laboratory tests | Throughout study
Plasma drug concentration versus time curve [AUC (0-t), AUC [0-∞], AUC(0-t)], maximum Cmax, tmax, and t1/2 of GSK1140115 as data permit | Duration of dosing

SECONDARY OUTCOMES:
Blood pressure (BP) and heart rate (HR) | Duration of dosing
Peak expiratory flow rate (PEFR) | Duration of Dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, Melbourne, Australia